CLINICAL TRIAL: NCT04598438
Title: Music to Enhance Auditory Encoding in Young Children: A Pilot Study
Brief Title: Music to Enhance Auditory Encoding in Young Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Patrick C. M. Wong, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Music_playgroup1
Record Dates: First submitted 2020-10-18; First posted 2020-10-22 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: Behavioral: Playgroup; Randomized Block Design; Therapy, Music; Parenting Education; Infant Development

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music intervention treatment group (Experimental): Participants attending the music behavioral early intervention program
  Interventions: Behavioral: Music behavioral early intervention program
- Arts and crafts active control group (Active Comparator): Participants attending the arts and crafts developmental enhancement program
  Interventions: Behavioral: Arts and crafts early enhancement program

INTERVENTIONS:
Behavioral: Music behavioral early intervention program — The program consists of carefully designed play-based enhancement strategies implemented in the form of hybrid online/in-person playgroups. Following a teach-model-coach-review approach, parents will learn to implement various skills that are expected to enhance infant's language and communication skills through singing and engaging in musical play with their child at home.
  Arms: Music intervention treatment group
Behavioral: Arts and crafts early enhancement program — The program follows the same general structure with the music intervention program. Parents will learn how to implement a series of arts and crafts activities at home, with an aim to enhance infant's visual-perceptual, motor, and sensory integration development.
  Arms: Arts and crafts active control group

SUMMARY:
The current pilot randomized control trial (RCT) examines whether active music participation enhances the encoding of speech in the neural auditory system which in turn leads to better language development in infants and toddlers. Healthy children will be randomized into either the music intervention treatment group or the arts and crafts active control group. Before and after treatment period, neural speech encoding and language and communication skills will be assessed. It is hypothesized that music intervention leads to enhanced neural speech encoding and language development compared to arts and crafts active control.

DETAILED DESCRIPTION:
Auditory encoding enables accurate representation of incoming speech signals, and can be measured by neural phase-locking to the frequencies of the speech stimulus via the frequency following response (FFR) (e.g., Wong et al., 2007). FFR measures are associated with a range of language processes including speech (Thompson et al., 2019) and literacy (White-Schwoch et al., 2015). Music intervention can lead to an enhanced FFR and auditory encoding in older children with poor language ability (e.g., Kraus et al., 2014). We therefore hypothesize that music intervention prescribed to young children (infants and toddlers) can also enhance FFR which will in turn enhance language and communication skills.

Participants: Cantonese-learning children between 8 to 12 months of age and their caregivers will participate in this research. All should report to be born healthy with gestational age of at least 37 weeks and birth weight of at least 2500g. We will enroll 48 children who will be randomized into the treatment or active control group (50% in each group) via blocked randomized (The Concise Encyclopedia of Statistics, 2008). Informed consent will be obtained from each family.

General Procedures: Within 2 weeks before and after treatment, children and families will undergo assessment (see outcome measures). Treatment will last for 10 weeks in a hybrid online and in-person delivery mode (see treatment procedures).

Outcome Measures: Infants will undergo EEG testing using an EEG system to elicit two types of responses, each lasting up to 10 minutes: 1) auditory encoding while they listen to auditory stimuli (e.g., Wong et al., 2007) and 2) resting-state EEG (e.g., Wilkinson et al., 2020). We will follow published procedures to derive neurophysiological metrics from the FFR signals such as pitch strength for speech encoding, and EEG spectral power analysis for amplitude of frequency bands at rest. The entire protocol will last under 30 min. Behavioral measures will include the MacArthur-Bates Communicative Development Inventories (MCDI)-Cantonese version (Tardif & Fletcher, 2008).

Treatment Procedures: Both treatment (music) and active control (arts and crafts) groups will consist of 10 weeks of training to take place online and in-person, led by a trained instructor. In addition, home practice will be assigned. Both will consist of a set of prescribed activities and materials and songs (for music treatment). For music, parents will be taught to use songs to implement activities to promote the child's auditory skills. For arts and crafts, a series of activities will promote visual perception (color, shape) and motor skills and encourage art making. A teach-model-coach-review approach (Roberts et al., 2014) will be implemented, with an important goal of teaching parents to implement the play sessions at home. Each family is required to complete a set of prescribed home practice activities and provide evidence of completion. These home activities will allow them to implement what they learn in the child's natural home environment and will encourage them to continue the activities they learn even after the completion of the treatment period.

Data Analysis: For each outcome measure, we will conduct a group x time ANOVA and expect a significant interaction. Posthoc analysis will reveal a larger, positive change in outcome measures for the treatment group relative to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Full-term infants, and their caregivers
* From families where Cantonese is the dominant language

Exclusion Criteria:

* Infants reported to fail the hearing sensitivity screening
* Infants with mental or neuro-motor disabilities associated with atypical development (e.g. birth asphyxia; major injuries; hypoxic-ischemic injury; significant growth restriction, and other indications of neurological abnormalities

Max Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2025-03-16 (Estimated)

PRIMARY OUTCOMES:
FFR auditory encoding measures | Up to 1 year after intervention
  Cortical and subcortical frequency following responses bands. Neurophysiological metrics of FFR signals derived from published procedures of auditory-evoked EEG, such as pitch strength for speech encoding will be submitted to statistical analyses.
Language developmental outcomes | Up to 1 year after intervention
  The MacArthur-Bates Communicative Development Inventories (MCDI)-Cantonese version

SECONDARY OUTCOMES:
Resting-state EEG signals | Up to 1 year after intervention
  EEG frequency bands measured at the resting-state. Typical analyses for resting-state EEG, such as spectral power analysis for amplitude of frequency bands will be adopted.

OTHER OUTCOMES:
Parenting practices and child-parent interaction | Up to 1 year after intervention
  At each visit to the lab, caregivers and children may be asked to engage in several age-appropriate tasks, during which they may be videotaped. Specifically, there will be semi-structured free play time (i.e. Symbolic and Non-symbolic play), book reading and sharing, and cognitive tasks (e.g., solving puzzles) etc. A parental questionnaire will be used to obtain paternal, maternal, and caregiver socio-demographic data, their health and family history, parenting style, and other relevant information about the caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Chun Man Wong, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Wong PCM, Vuong LC, Liu K. Personalized learning: From neurogenetics of behaviors to designing optimal language training. Neuropsychologia. 2017 Apr;98:192-200. doi: 10.1016/j.neuropsychologia.2016.10.002. Epub 2016 Oct 5. PMID 27720749
- [Background] White-Schwoch T, Woodruff Carr K, Thompson EC, Anderson S, Nicol T, Bradlow AR, Zecker SG, Kraus N. Auditory Processing in Noise: A Preschool Biomarker for Literacy. PLoS Biol. 2015 Jul 14;13(7):e1002196. doi: 10.1371/journal.pbio.1002196. eCollection 2015 Jul. PMID 26172057
- [Background] Thompson EC, Krizman J, White-Schwoch T, Nicol T, Estabrook R, Kraus N. Neurophysiological, linguistic, and cognitive predictors of children's ability to perceive speech in noise. Dev Cogn Neurosci. 2019 Oct;39:100672. doi: 10.1016/j.dcn.2019.100672. Epub 2019 Aug 6. PMID 31430627
- [Background] Kraus N, Slater J, Thompson EC, Hornickel J, Strait DL, Nicol T, White-Schwoch T. Music enrichment programs improve the neural encoding of speech in at-risk children. J Neurosci. 2014 Sep 3;34(36):11913-8. doi: 10.1523/JNEUROSCI.1881-14.2014. PMID 25186739
- [Background] Wilkinson CL, Gabard-Durnam LJ, Kapur K, Tager-Flusberg H, Levin AR, Nelson CA. Use of longitudinal EEG measures in estimating language development in infants with and without familial risk for autism spectrum disorder. Neurobiol Lang (Camb). 2020;1(1):33-53. doi: 10.1162/nol_a_00002. Epub 2020 Apr 6. PMID 32656537
- [Background] Tardif, T., Fletcher, P., Zhang, Z. X., Liang, W. L., Zuo, Q. H., & Chen, P. (2008). User's guide and manual for the Chinese communicative development inventories (Putonghua and Cantonese). Beijing, China: Peking University Medical Press.
- [Background] Roberts MY, Kaiser AP, Wolfe CE, Bryant JD, Spidalieri AM. Effects of the teach-model-coach-review instructional approach on caregiver use of language support strategies and children's expressive language skills. J Speech Lang Hear Res. 2014 Oct;57(5):1851-69. doi: 10.1044/2014_JSLHR-L-13-0113. PMID 24950492
- [Background] (2008) Randomized Block Design. In: The Concise Encyclopedia of Statistics. Springer, New York, NY. https://doi.org/10.1007/978-0-387-32833-1_344